CLINICAL TRIAL: NCT06003062
Title: Suppression of Upper Lip Hair Growth Using Novel Hemp Extract - A Case Series
Brief Title: Suppression of Upper Lip Hair Growth Using Novel Hemp Extract
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical Life Care Planners, LLC (Other)
Responsible Party: Principal Investigator, Gregory L Smith, MD, MPH, Principal Investigaor, Medical Life Care Planners, LLC
Other Study IDs: Lip Hair Growth Suppression
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hirsutism; Hair Diseases
Keywords: Narcissus Tarzetta Bulb Extract; Cannabinoid One (CB1) receptor; IBR-Dormin; Hemp-extract
MeSH Terms: conditions — Hirsutism; Hair Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard Topical NIghtly Dose: Treatment group
  Interventions: Drug: Narcissus Tazetta Bulb Extract and Novel Hemp Extract

INTERVENTIONS:
Drug: Narcissus Tazetta Bulb Extract and Novel Hemp Extract — Topical nightly application of phytonutraceutical

SUMMARY:
A clinical case series will be conducted measuring upper lip hair suppression for cosmetic effects in a group of 25 adult women with hirsutism of the upper lip. The study will use a topical phytonutraceutical that contains two ingredients that have been shown to suppress hair growth. The serum contains Narcissus Tazetta Bulb Extract (0.2%) and a hemp-extract (0.15%) known to stimulate cannabinoid one (CB1) receptors.

The subjects will use the serum nightly for 60 days. High-power ProScope photographs will be obtained at the philtrum (above the center of the upper lip) as a landmark. Prior to starting the serum subjects will grow their upper lip hair for seven days. Hair shafts will be counted and graded for thickness and color using a standard methodology. The subjects will then use the serum for 60 days and will not be allowed to use laser, waxing, bleaching or tweezing during the duration of the study. Only shaving will be allowed. At the end of the 60 day course the subjects will grow their lip hair for seven days and the high-power photographs will be repeated at the same location based on landmarks.

An independent board-certified dermatologist will evaluate and grade the pre- and post- serum photographs for cosmetic effects, number and thickness of the hairs.

DETAILED DESCRIPTION:
Hirsutism is defined as increased bodily and facial hair growth in females presenting in locations where hair is ordinarily minimal or absent. It affects almost 30% of adult females during their lifetime. Current treatments for hirsutism include the use of oral contraceptives or antiandrogens. These drugs and hormones are associated with adverse effects and they may not manifest results if at all for at least 6 months most cannot be used if the female is pregnant, breastfeeding, or trying to become pregnant. Many women find that a multipronged approach that includes direct hair removal (such as plucking, waxing, shaving, depilatories, bleaches and laser), suppression of androgen production with drugs. More recently an effective prescription topical cream, Eflornithine hydrochloride (brand name: Vaniqa) has become available to slow the growth of unwanted facial hair in women. It does not remove hair permanently. Noticeable results take approximately six to eight weeks, and once the cream is discontinued, hair returns to pretreatment levels after approximately eight weeks. Eflornithine cream may cause skin to redden.

Narcissus Tarzetta Bulb Extract 0.02% IBR-Dormin applied topically reduced hair shaft elongation by 34%. The test also showed the hair follicle started the transition from growth to resting phase (telogen). A study of 3.0% topical extract revealed a delay of men's facial hair regrowth after shaving.

Studies of endocannabinoids and phytocannabinoids that stimulate the cannabinoid one (CB1) receptor reveal that topical application inhibited hair shaft elongation and the proliferation of hair matrix keratinocytes, and induced intraepithelial apoptosis and premature hair follicle regression (catagen).

A clinical case series from serial patients with hirsuitism (adult females) at a dermatology clinic will be conducted measuring upper lip hair suppression for cosmetic effects and change in hair shaft count and color. The study will use a topical phytonutraceutical containing Narcissus Tazetta Bulb Extract (0.2%) and a hemp-extract (0.15%) known to stimulate cannabinoid one (CB1) receptors. Based on prior studies the topical will work locally as a locally active topical without systemic absorption.

The 25 subjects will use the serum nightly for 60 days. High-power ProScope photographs will be obtained at the philtrum (above the center of the upper lip) as a landmark. Prior to starting the serum subjects will grow their upper lip hair for seven days. Hair shafts will be counted and graded for thickness and color using a standard methodology. The subjects will then use the serum for 60 days and will not be allowed to use laser, waxing, depilatories, bleaching or tweezing during the duration of the study. Only shaving will be allowed. At the end of the 60-day trial the subjects will grow their lip hair for seven days and the high-power photographs will be repeated at the same location based on landmarks.

An independent board-certified dermatologist will evaluate and grade the pre- and post-treatment photographs for cosmetic effects, number and thickness of the hairs.

ELIGIBILITY:
Inclusion Criteria:

Physician diagnosed upper lip hirsutism Prior use of therapies to treat the upper lip hirsutism No laser, depilation, or waxing within prior 8 weeks -

Exclusion Criteria:

Local infection near or at application site. Local skin irritation or ulceration near or at application site. Inability to be available for entire duration of study and in-person photographs

-

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women
Study Population: Adult women with physician-diagnosed hirsutism presenting to a dermatology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Hair Follicle Number | 60 days
  The change in the number of identifable hair follicles using high-power ProScope
Hair Follicle Diameter | 60 days
  The change in the hair average hair follicle diameter using high-power ProScope

SECONDARY OUTCOMES:
Hair Shaft Color | 60 days
  The change in the darkness of the hair follicles will be measured using high-power ProScope

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kopera D, Wehr E, Obermayer-Pietsch B. Endocrinology of hirsutism. Int J Trichology. 2010 Jan;2(1):30-5. doi: 10.4103/0974-7753.66910. PMID 21188021
- [Background] Gupta AK, Talukder M. Cannabinoids for skin diseases and hair regrowth. J Cosmet Dermatol. 2021 Sep;20(9):2703-2711. doi: 10.1111/jocd.14352. Epub 2021 Aug 7. PMID 34363728
- [Background] Barrionuevo P, Nabhan M, Altayar O, Wang Z, Erwin PJ, Asi N, Martin KA, Murad MH. Treatment Options for Hirsutism: A Systematic Review and Network Meta-Analysis. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1258-1264. doi: 10.1210/jc.2017-02052. PMID 29522176